CLINICAL TRIAL: NCT01137630
Title: A Multicenter, Randomised Double Blind, Placebo Controlled Study of Efficacy, Safety and Tolerability of Two Topical K40 Formulations in Adults With Seborrhoeic Dermatitis (SD) of the Scalp.
Brief Title: Two Topical K40 Formulations in Adults With Seborrhoeic Dermatitis (SD) of the Scalp
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Moberg Pharma AB (Industry)
Responsible Party: Kjell Rensfeldt MD, Moberg Derma AB
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K40-3
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2010-06

CONDITIONS: Seborrhoeic Dermatitis of the Scalp
Keywords: seborrhoeic dermatitis; scalp; K40a; K40b
MeSH Terms: conditions — Dermatitis, Seborrheic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- K40a (Experimental): K40a is to be applied to affected areas of the scalp once daily for 4 weeks. Thereafter, a maintenance phase of 4 weeks is to follow with application 3 times per week. Approximately one tablespoon of the respective formulation is to be applied before bed and to be washed out with the patient's normal shampoo in the morning.
  Interventions: Drug: K40a
- K40b (Experimental): K40b is to be applied to affected areas of the scalp once daily for 4 weeks. Thereafter, a maintenance phase of 4 weeks is to follow with application 3 times per week. Approximately one tablespoon of the respective formulation is to be applied before bed and to be washed out with the patient's normal shampoo in the morning.
  Interventions: Drug: K40b
- Placebo (Placebo Comparator): Placebo is to be applied to affected areas of the scalp once daily for 4 weeks. Thereafter, a maintenance phase of 4 weeks is to follow with application 3 times per week. Approximately one tablespoon of the respective formulation is to be applied before bed and to be washed out with the patient's normal shampoo in the morning.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: K40a — One tablespoon is to be applied to affected areas of the scalp once daily for 4 weeks. Thereafter, a maintenance phase of 4 weeks is to follow with application 3 times per week.
  Other Names: K301a
  Arms: K40a
Drug: K40b — One tablespoon is to be applied to affected areas of the scalp once daily for 4 weeks. Thereafter, a maintenance phase of 4 weeks is to follow with application 3 times per week.
  Arms: K40b
Drug: Placebo — One tablespoon is to be applied to affected areas of the scalp once daily for 4 weeks. Thereafter, a maintenance phase of 4 weeks is to follow with application 3 times per week.
  Arms: Placebo

SUMMARY:
Seborrhoeic dermatitis (SD) is a papulosquamous (presence of both papules and scales) disorder patterned on the sebum-rich areas of the scalp, face, and trunk.

The current treatment does not cure the disease permanently. Therefore it must be repeated when the symptoms recur, or even prophylactically. Corticosteroids and antifungals are the mainstay of therapy. Topical corticosteroids rapidly reduce the cutaneous signs of disease, but are associated with a high frequency of relapse when treatment is stopped. They are reserved for acute flare-ups only as they may precipitate recurrences and dependence. In addition, chronic use of corticosteroids is associated with side-effects.

The scientific rationale for the use of K40 for treatment of SD was based on clinical evidence that K40 improves erythema and desquamation with mild adverse reactions in a few cases. The primary objective of the study was to evaluate the efficacy of K40 (K40a and K40b combined) compared to placebo after 4 weeks treatment as measured by the sum of erythema and desquamation scores at Week 4.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (including fertile women)
* 18-65 years of age
* Seborrhoeic dermatitis of the scalp for at least 2 months
* Presenting erythema and desquamation of mild, moderate, pronounced or severe intensity
* Signed written informed consent

Exclusion Criteria:

* Patient on an antifungal, selenium sulphite or corticosteroid therapy within the last 2 weeks prior to start of study treatment
* Any other cutaneous disease of the face requiring a specific topical treatment (corticosteroids, antifungals, antibiotics, retinoids, benzoyl peroxide or a-hydroxyacids) during the previous 15 days
* Oral treatment with cyclines, lithium, antifungals or inhaled corticosteroids during the previous month
* Use of systemic corticosteroids and retinoids during the previous 2 months
* SD associated with Parkinson's disease, human immunodeficiency virus infection
* Current or any history of ear, nose and throat carcinoma,
* Current or any history of severe concomitant disease according to Investigator'sjudgement
* Allergy to any of the tested treatment components

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2007-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Erythema and desquamation scores | Week 4
  Sum of erythema and desquamation scores at Week 4

SECONDARY OUTCOMES:
Erythema and desquamation scores | Weeks 2 and 8
  Sum of erythema and desquamation scores at Week 2 and 8
Responder | Weeks 2, 4 and 8
  Responder defined as a patient with complete remission (sum of erythema and desquamation scores=0) or partial remission (sum of scores=1 or 2) at Week 2, 4 and 8
Erythema score | Weeks 2, 4 and 8
  Erythema score at Week 2, 4 and 8
Desquamation score | Weeks 2, 4 and 8
  Desquamation score at Week 2, 4 and 8
Doctor's Global evaluation | Week 4 and 8
  Doctor's Global evaluation at Week 4 and 8
Patient's Global evaluation | Weeks 4 and 8
  Patient's Global evaluation at Week 4 and 8
Pruritus score | Weeks 2, 4 and 8
  Patient's pruritus score at Week 2, 4 and 8
Dandruff score | Weeks 2, 4 and 8
  Patient's dandruff score at Week 2, 4 and 8
Dermatology Life Quality Index | Week 4 and 8
  Dermatology Life Quality Index (DLQI) assessed by the patient at Week 4 and 8
Ease of application | Weeks 4 and 8
  Cosmetic properties; ease of application at Week 4 and 8
Stickiness | Weeks 4 and 8
  Cosmetic properties; stickiness at Week 4 and 8
Effect on hair quality | Weeks 4 and 8
  Cosmetic properties; effect on hair quality at Week 4 and 8
Adverse events | Weeks 0, 2, 4 and 8
  Adverse Events classified by body system and preferred term

CONTACTS AND LOCATIONS:
Overall Officials: Lennart Emtestam, MD, Principal Investigator — Karolinska University Hospital
Locations (11):
- Sweden (11):
  - Dellenkliniken, Delsbo
  - Läkarhuset Farsta Centrum, Farsta
  - Stortorgets Hälsocentral, Gävle
  - Hedesunda Hälsocentral, Hedesunda
  - Familjehälsan, Hofors
  - Derbykliniken, Malmo
  - Möllevångens Läkargrupp,, Malmo
  - Möllevångens Läkargrupp, Malmo
  - Österpraktiken, Örebro
  - Department of Dermatology, Karolinska University Hospital, Stockholm
  - Hälsojouren, Uppsala